CLINICAL TRIAL: NCT04079595
Title: Randomized Controlled Trial Comparing Closed vs. Open Face Masks for Cranial Radiotherapy
Brief Title: Closed vs. Open Face Masks for Cranial Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Comfort RCT
Record Dates: First submitted 2019-07-11; First posted 2019-09-06 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Brain Tumor; Brain Metastases; Small Cell Lung Cancer; Meningioma
MeSH Terms: conditions — Brain Neoplasms; Small Cell Lung Carcinoma; Meningioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open-faced head immonbilization masks (Experimental): Masks used for immobilization of the head (CIVCO Radiotherapy, Orange City, Iowa) during radiation therapy with openings for the face
  Interventions: Device: Head immobilization mask
- Closed-face head immobilization masks (Active Comparator): Masks used for immobilization of the head (CIVCO Radiotherapy, Orange City, Iowa) during radiation therapy with the face closed
  Interventions: Device: Head immobilization mask

INTERVENTIONS:
Device: Head immobilization mask — Immobilization

SUMMARY:
The aim of the study is to evaluate whether open-face masks improve patient comfort/preference whilst maintaining immobilization performance as known for closed masks in patients undergoing whole or partial cranial radiotherapy.

DETAILED DESCRIPTION:
Upon randomization, patients will be begin treatment either with an open-face mask (A) or closed mask (B). Two individual immobilization masks - the open-face and closed masks - will be fabricated for every single patient. During the 1st half of treatment the randomly assigned mask will be used followed by using another mask for the 2nd half of treatment. Discomfort/pain/anxiety and mask preference will be scored during treatment with a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and International Council for Harmonization (ICH)/Good Clinical Practice (GCP) regulations before any trial specific procedures;
* Indication for cranial radiotherapy irrespective of tumor type;
* Age: ≥ 18 years old;
* Karnofsky performance status ≥70;
* Patients who are willing and able to comply with scheduled visits, treatment, and other trial procedures.

Exclusion Criteria:

* Cranial radiotherapy in less than 10 fractions;
* Prior brain irradiation;
* Inability to complete magnetic resonance imaging (MRI) procedure due to claustrophobic anxiety;
* Women who are pregnant or breast feeding;
* Intention to become pregnant during the course of the trial;
* Lack of safe contraception;
* Known or suspected non-compliance, drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Patient discomfort with the two immobilization masks | Change in patient discomfort through the course of radiation therapy, up to 6 weeks
  Patient discomfort measured with the Visual Analogue Scale (VAS) 0-10 with "no discomfort" (scored as 0) and "extreme discomfort" (scored as 10).
Mask preference | At completion of radiation therapy, up to 6 weeks depending on radiation dose fractionation
  Mask preference measured with the Yes/No questionnaire. Upon completion of radiation therapy patients will be asked which of the two immobilization masks they prefer - either Yes or No to one of the used masks.

SECONDARY OUTCOMES:
Treatment set-up accuracy | Through the course of radiation therapy, up to 6 weeks
  Measured with planar kilovoltage (kV) imaging
Treatment intra-fraction accuracy | Through the course of radiation therapy, up to 6 weeks
  Measured with an optic surface imaging (OSI) system
Immobilization-mask-induced severe adverse events during treatment | From the baseline to 3 months post-treatment
  Measured with CTCAE version 5.0
Location of discomfort on the head/face | Changes in location of discomfort on the head/face through the course of radiation therapy up to 6 weeks
  Measured with the questionnaire consisting of a head/face diagram divided in 8 regions

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Guckenberger, Dr., Principal Investigator — University Hospital Zurich, Department of Radiation Oncology
Locations (1):
- Department of Radiation Oncology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Randomized self-controlled study comparing open-face vs. closed immobilization masks in fractionated cranial radiotherapy — https://pubmed.ncbi.nlm.nih.gov/38677329/